CLINICAL TRIAL: NCT02634203
Title: Riociguat Versus Balloon Pulmonary Angioplasty in Non-operable Chronic thromboEmbolic Pulmonary Hypertension
Acronym: RACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOM14123; 2015-A00973-46 (Other: IDRCB)
Record Dates: First submitted 2015-12-08; First posted 2015-12-17 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2017-11

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: Chronic Thromboembolic Pulmonary Hypertension; Balloon Pulmonary Angioplasty; Riociguat
MeSH Terms: interventions — riociguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Balloon Pulmonary Angioplasty (BPA) (Experimental): Non-operable patients with CTEPH allocated to BPA arm
  Interventions: Procedure: Balloon Pulmonary Angioplasty (BPA)
- Riociguat (Active Comparator): Non-operable patients with CTEPH allocated to Riociguat arm
  Interventions: Drug: Riociguat

INTERVENTIONS:
Procedure: Balloon Pulmonary Angioplasty (BPA) — Balloon pulmonary angioplasty (BPA) will be done via femoral vein. 2 sessions will be performed during the same hospitalization following by additional sessions at an interval of 2-3 weeks until a mean PAP< 30 mmHg is achieved A pulmonary angiography and a right heart catheterization will be performed at each BPA session
  Arms: Balloon Pulmonary Angioplasty (BPA)
Drug: Riociguat — The starting dose will be 1 mg three times daily as recommended. The dose will be titrated every 2 weeks according to the peripheral systolic pressure. Dose should be increased by 0.5 mg three times daily every two weeks to a maximum of 2.5 mg three times daily, if systolic blood pressure is ≥95 mmHg and the patient has no signs or symptoms of hypotension.
  Other Names: Medical therapy with Riociguat
  Arms: Riociguat

SUMMARY:
"Chronic thromboembolic pulmonary hypertension (CTEPH) is a severe form of pulmonary hypertension characterized by obstruction of the pulmonary vasculature by residual organized thrombi, leading to increased pulmonary vascular resistance (PVR), progressive pulmonary hypertension, and right failure.

In patients deemed operable, pulmonary endarterectomy (PEA) is the gold standard treatment and is the only potentially curative treatment. However, some patients are ineligible for surgery owing to occlusion of distal vessels. The best treatment option for these non-operable CTEPH patients is not yet established.

DETAILED DESCRIPTION:
Currently, riociguat is the only drug approved in Europe and US for the treatment of non-operable CTEPH. However, medical therapy with riociguat does not address obstructive lesions. In this sense, another treatment option, balloon pulmonary angioplasty (BPA), began recently to gain widespread interest after development in several centers. This procedure uses the standard balloon angioplasty technique to dilate selected pulmonary arteries. The main aim is to reopen vessels occluded by webs and bands. Several teams, mainly from Japan, have reported their experiences with BPA for the treatment of non-operable CTEPH and demonstrated impressive decrease in pulmonary vascular resistance and improvement in functional status and exercise capacity with an acceptable procedure-related risk. Although BPA has never been prospectively evaluated, most of the leading CTEPH centers worldwide have currently added BPA to their therapeutic options. However, no randomized controlled trial comparing safety and efficacy of medical therapy with riociguat versus pulmonary balloon angioplasty has been performed so far. Therefore, the respective places of medical treatment and of BPA in the management of inoperable patients with CTEPH need to be further evaluated.

An ancillary study will evaluate the efficacy and safety of employment of two sequentially used treatments at 12 months. The studied population is that of the study RACE. The patient follow-up period will be extended by 6 months, its duration of participation will be in total of 13 months. The exams will be the same as those of the V3 of the RACE study.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years of age at Visit 1
* CTEPH patients considered as non-operable but eligible for balloon pulmonary angioplasty and riociguat by the multidisciplinary meeting, with pulmonary vascular resistance > 320 dyn.sec.cm-5 and mean PAP > 25 mmHg and PWP (Pulmonary capillary Wedge Pressure) ≤ 15 mmHg measured at least 3 months after start of full anticoagulation. If the patient is treated with new oral anticoagulants drugs, NOAC's, (rivaroxaban, apixaban, dabigatran), the treatment should be switched to Vitamin K antagonist (VKA).
* The diagnosis of CTEPH must have been established based on 2 of the 3 following methods before study entry: ventilation-perfusion scan, pulmonary angiography, spiral-CT scan.
* The diagnosis of inoperability must have been established based on spiral-CT scan and/or pulmonary angiography before study entry.
* Unspecific treatments which may also be used for the treatment of pulmonary hypertension (PH) such as oral anticoagulants, diuretics, digitalis, calcium channel blockers or oxygen supplementation are permitted. However treatment with anticoagulants must have been started at least 3 months before Visit 1.
* Specific PH treatments (bosentan, ambrisentan, macitentan, sildenafil, tadalafil, epoprostenol, treprostinil, iloprost) are not permitted at Visit 1.
* Patients who fulfill criteria for a supplemental long-term oxygen therapy (PaO2 < 55 mmHg at rest) need to be supplied sufficiently before study entry. The amount of supplemental oxygen and the delivery method need to be stable for at least one month before Visit 1.
* Right-heart catheterization results for the definite diagnosis of PH must not be older than 6 weeks at Visit 1 (will be considered as baseline values), must have been measured after at least 3 months of full anticoagulation, and must have been measured in the participating center under standardized conditions.
* Women without childbearing potential defined as postmenopausal women aged 55 years or older, women with bilateral tubal ligation, women with bilateral ovarectomy, and women with hysterectomy can be included in the study. Women with childbearing potential can be included in the study only if a serological pregnancy test is negative and a combination of condoms with a safe and highly effective contraception method is used.
* Patients who are able to understand and follow instructions and who are able to participate in the study for the entire period.
* Patients must have given their written informed consent to participate in the study after having received adequate previous information and prior to any study-specific procedures.

Exclusion Criteria:

* Participation in another clinical trial during the preceding 3 months.
* Pregnant women, or breast feeding women, or women with childbearing potential not using a combination of condoms and a safe and highly effective contraception method (hormonal contraception with implants or oral contraceptives, intrauterine devices ).
* Patients with a medical disorder, condition, or history of such that would impair the patient's ability to participate or complete this study in the opinion of the investigator.
* Patients with underlying medical disorders and anticipated life expectancy below 2 years (eg active cancer disease with localized and/or metastasized tumor mass).
* Patients with a history of severe allergic-like reaction to intravascular administration of iodinated contrast media (including diffuse edema or facial edema with dyspnea, diffuse erythema with hypotension, laryngeal edema with stridor and/or hypoxia, bronchospasm, anaphylactic shock with hypotension and tachycardia)
* Significant obstructive or restrictive lung disease (forced expiratory volume < 60% predicted and/or total lung capacity < 70% predicted).
* Severe hepatic impairment (Child-Pugh C)
* Left heart failure with an ejection fraction less than 40%
* Severe proven or suspected coronary artery disease (symptomatic patients with Canadian Cardiovascular Society Angina Classification class 2-4, and/or requiring nitrates, and/or myocardial infarction within the last 3 months before Visit 1).
* Severe renal insufficiency (glomerular filtration rate ≤ 30mL/min eg calculated based on the Cockcroft formula).
* Patient not covered by social security service

Non-inclusion criteria related to treatment by riociguat:

* Patients with significant interstitial lung disease on High-resolution computed tomography (HRCT)
* Patients with hypersensitivity to riociguat or any of the excipients.
* Treatment with :

  * PDE-5 Inhibitors (eg Sildenafil or Tadalafil)
  * NO donors (eg Nitrates)
* Strong multi pathway cytochrome P450 (CYP) and P-glycoprotein (P-gp) / breast cancer resistance protein (BCRP) inhibitors such as azole antimycotics (e.g. ketoconazole, itraconazole) or HIV protease inhibitors (e.g. ritonavir)
* Systolic blood pressure <95mmHg
* Patients with a history of life-threatening hemoptysis (>100 mL in 24 h) or who have previously undergone bronchial arterial embolization for hemoptysis

Non-inclusion criteria related to BPA:

• Patients who could not remain in a supine position for at least 120 min for any reason.

Very distal CTEPH disease without stenosis, webs, or slits on CT scan and CTEPH disease with predominant complete occlusions of segmental or sub- segmental arteries (defined by the multidisciplinary meeting)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Pulmonary Vascular Resistance (PVR) | Baseline and at 26 weeks
  Pulmonary Vascular Resistance (PVR)

SECONDARY OUTCOMES:
Change from Baseline in 6 Minute Walking Distance (6MWD) | Baseline and at 26 weeks
  6 Minute Walking Distance (6MWD)
Change from Baseline in WHO (World Health Organization) functional class (FC) | Baseline and at 26 weeks
  WHO functional class (FC)
Change from baseline in NT PRO-BNP | Baseline and at 26 weeks
  NT PRO-BNP (N Terminale Pro-Brain Natriuretic Peptide ) results
Change from Baseline in Borg dyspnea score (measured at the end of the 6MWD Test | Baseline and at 26 weeks
  Borg dyspnea score (measured at the end of the 6MWD Test)
Time To Clinical Worsening defined by the occurence of - Death (all-cause mortality or Lung) - or Heart-lung transplantation - or Hospitalization due to persistent worsening of PH or - Start of PAH specific treatment | Up to 26 weeks
  Clinical Worsening

CONTACTS AND LOCATIONS:
Overall Officials: Xavier JAIS, MD, PhDI, Principal Investigator — AP-HP, Bicêtre Hospital
Locations (1):
- AP-HP, Bicêtre Hospital, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gerges C, Jevnikar M, Brenot P, Savale L, Beurnier A, Bouvaist H, Sitbon O, Fadel E, Boucly A, Chemla D, Simonneau G, Humbert M, Montani D, Jais X; RACE Investigators. Effect of Balloon Pulmonary Angioplasty and Riociguat on Right Ventricular Afterload and Function in CTEPH: Insights From the RACE Trial. Circ Cardiovasc Interv. 2025 Feb;18(2):e014785. doi: 10.1161/CIRCINTERVENTIONS.124.014785. Epub 2025 Feb 18. PMID 39965044
- [Derived] Jais X, Brenot P, Bouvaist H, Jevnikar M, Canuet M, Chabanne C, Chaouat A, Cottin V, De Groote P, Favrolt N, Horeau-Langlard D, Magro P, Savale L, Prevot G, Renard S, Sitbon O, Parent F, Tresorier R, Tromeur C, Piedvache C, Grimaldi L, Fadel E, Montani D, Humbert M, Simonneau G. Balloon pulmonary angioplasty versus riociguat for the treatment of inoperable chronic thromboembolic pulmonary hypertension (RACE): a multicentre, phase 3, open-label, randomised controlled trial and ancillary follow-up study. Lancet Respir Med. 2022 Oct;10(10):961-971. doi: 10.1016/S2213-2600(22)00214-4. Epub 2022 Aug 1. PMID 35926542